CLINICAL TRIAL: NCT00368160
Title: The Effects of a Single Evening Dose of 3 mg Eszopiclone on Next Day Driving Ability and Psychomotor/Memory Function in Healthy Volunteers Compared to Placebo
Brief Title: Study of an Evening Dose of Eszopiclone on Next Day Driving Ability & Psychomotor/Memory Function in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-059
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: Next day driving
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): eszopiclone 3 mg
  Interventions: Drug: Eszopiclone
- 2 (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — eszopiclone 3 mg
  Other Names: S-Zopiclone; Lunesta
  Arms: 1
Drug: Placebo — Placebo tablet
  Arms: 2

SUMMARY:
Male and female healthy volunteers. Patients must also possess a full current driving license (for at least one year), and be a regular car driver.

DETAILED DESCRIPTION:
The study is a single centre, randomised, double blind, placebo controlled 2-way crossover design in a group of 32 healthy male and female volunteers. The medications under investigation are eszopiclone and placebo. Volunteers will receive the study medications and placebo on the evening of Day 2 of each treatment period. Performance will be assessed on Day 3 of each treatment period. Each treatment period will be separated by at least a 7-day washout period. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55 years inclusive
* In good health as determined by a medical history, ECG, haematology, blood and urine biochemistry and physical examination by the doctor
* A body mass index greater than or equal to 18 and less than or equal to 30
* Registered with a general practitioner (GP)
* Hold a full current driving licence for at least one year, and be regular car drivers

Exclusion Criteria

* Clinically significant use of psychotropic medication in the last three months. For example, this would include the prolonged use of antidepressants, antipsychotics, or antihistamines, but would exclude the occasional use of cold or flu remedies (which often contain antihistamines and/ or opiates)
* The use of any other medication in the last two weeks with the exception of oral, transdermal, IUDs (progestogen only contraceptive e.g. Mirena), or depot contraceptives, non-steroidal analgesics (e.g. ibuprofen), and paracetamol
* Significant history of mental illness, significant drug allergy, malignancy or chronic drug abuse (including alcohol)
* Any subject with known hypersensitivity to any of the study treatments
* A sleep/ wake cycle (e.g. shift work) liable to prejudice the results of the study
* Pregnant or lactating females, and females of child bearing potential not using effective contraception
* Volunteers who habitually smoke more than 5 cigarettes per day
* Caffeine consumption of more than 5 cups or glasses per day
* History of alcohol or drug dependence or intake of more than the equivalent of 14 units of alcohol per week for females and 21 units per week for males
* Current participation in another clinical trial, or participation in a clinical trial within the last 90 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
next day performance in a standardised test of car driving | 9.5 hours post dose

SECONDARY OUTCOMES:
Compensatory Tracking Task (CTT) | 9.5 hours post dose
Rapid Visual Information Processing (RVIP) | 9.5 hours post dose
Sternberg's Short-term Memory Scanning task (STM) | 9.5 hours post dose
Critical Flicker Fusion (CFF) | 9.5 hours post dose
Digit Symbol Substitution Test (DSST) | 9.5 hours post dose
Choice Reaction Time (CRT) | 9.5 hours post dose
Leeds Sleep Evaluation Questionnaire and Leeds Analogue Rating Scales | 9.5 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- HPRU Medical Research Centre, Guildford, Surrey, United Kingdom